CLINICAL TRIAL: NCT05497076
Title: A Single-center, Single-arm, Phase Ib Clinical Study of the Efficacy and Safety of Dalpiciclib Combined With Third-generation EGFR-TKI in Patients With EGFR Mutation and Meningial Metastasis in Non-small Cell Lung Cancer Progressing Through Third-generation TKI and Platinum-containing Two-drug Chemotherapy
Brief Title: the Efficacy and Safety of Dalpiciclib Combined With Third-generation EGFR-TKI in Patients With EGFR Mutation and Meningial Metastasis in Non-small Cell Lung Cancer Progressing Through Third-generation TKI and Platinum-containing Two-drug Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: LM20220606
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Non-small Cell Lung Cancer Confirmed by Histopathology or Cytology; The TNM (8th) Phase is IV; With EGFR Mutations; Meningeal Progression Occurred After Previous Platinum-containing Two-drug Chemotherapy and Third-generation EGFR-TKI Treatment; Male or Female; The Age of 18 Years Old or More; ECOG PS 0 to 2 Points

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Efficacy and safety of Dalpiciclib combined with third-generation EGFR-TKI in patients with advanced EGFR-mutated non-small cell lung cancer with meningeal metastasis after third-generation TKI and platinum-containing chemotherapy

DETAILED DESCRIPTION:
Subjects with advanced NSCLC who developed meningeal progression after previous platinum-based two-drug chemotherapy and third-generation EGFR-TKI treatment were enrolled.

Exploratory analysis: Peripheral blood and/or cerebrospinal fluid samples were retained before medication, 4 weeks after medication, and after progression. Cdk4/6, CDKN2A, CDKN2B, CCND1 (Cyclin D1), CCND2 (Cyclin D2) and CCND3 (Cyclin D2) were detected by NGS D3), CCNE1, RB1 cell cycle pathway changes and subjects without these changes in stratification, namely whether the above cell cycle regulation abnormalities can be used as biomarkers for efficacy prediction and prognosis. And whether there are differences in the expression of the above genes in peripheral blood and cerebrospinal fluid, to explore the relationship between intracranial and extracranial cell cycle regulation abnormalities in the upstream and downstream pathways.

The first stage was the safety introduction period, in which the previous drugs and fixed doses of the third generation EGFR-TKI were continued, and Dalpiciclib was enrolled in the 3+3 mode. After one subject was enrolled, the second subject was enrolled after completing the dose-limiting toxicity (DLT) observation period (3 weeks). If no DLT was found in the 3 subjects, the next dose ramp could be performed. If there was 1 DLT, 3 patients of this dose grade were added to the group. If no DLT was found in any of the 3 cases, the next dose grade was entered. It is planned to enroll 6 to 9 subjects. According to the safety data obtained during the safety observation period, it will be determined whether to add other dose groups for exploration in the first stage after comprehensive analysis and discussion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 when signing informed consent, both male and female;
2. Advanced or metastatic NSCLC confirmed by histology or cytology is stage IV according to THE TNM stage of lung cancer, IASLC 2015 Eighth Edition;
3. EgFR-sensitive mutations (exon 19 deletion, exon 21 L858R or L861Q mutation, exon 18 G719X mutation, etc.) exist. Meningeal progression follows platinum-containing chemotherapy in combination with/without antivascular and/or in combination with/without immunotherapy, and 3 generations of EGFR-TKI (which can be 1+3, 2+3 or directly after 3 generations of targeted therapy). Patients with BMS can be treated with brain radiotherapy. Cerebrospinal fluid and peripheral blood were collected for EXPLORATORY NGS testing. Subjects identified with cdK4/6, CDKN2A, CDKN2B, CCND1 (Cyclin D1), CCND2 (Cyclin D2), CCND3 (Cyclin D3), CCNE1 and RB1 cell cycle pathway changes by genetic testing were stratified for analysis;
4. ECOG PS score: 0-2;
5. Normal function of major organs, that is, meeting the following criteria: a) blood routine examination (no blood transfusion within 14 days, no hematopoietic stimulation drugs correction) : Hemoglobin (Hb) ≥90g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet (PLT) ≥100×109/L; White blood cell count (WBC) ≥3.0×109/L; B) Biochemical examination: ALT and AST ≤2.5× upper limit of normal value (ULN); Serum total bilirubin (TBIL) ≤1.5×ULN; Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥50ml/min; If liver metastasis was present, total bilirubin ≤3×ULN, ALT and AST≤5×ULN; C) Coagulation function: activated partial thrombin time (APTT), international standardized ratio (INR), prothrombin time (PT) ≤1.5×ULN; D) Doppler ultrasound assessment: left ventricular ejection fraction (LVEF)≥50%;
6. a washout period of at least 21 days between the last dose of chemotherapy and enrollment (if the patient did not receive radiotherapy); Patients undergoing brain radiation therapy must complete and fully recover from the acute toxicity of radiation therapy. A washout period of at least 14 days is required between the end of radiotherapy and enrollment.
7. The expected survival time is not less than 3 months;
8. Allow asymptomatic BMS who are stable and do not require steroid treatment for more than 4 weeks before the study begins;
9. Patient can swallow oral medication;
10. Women of childbearing age must have a negative pregnancy test (serum or urine) within 14 days prior to enrollment and voluntarily use an appropriate method of contraception during the observation period and within 3 months after the last administration of the study drug; For men, surgical sterilization or consent to use appropriate methods of contraception during the observation period and for 3 months after the last administration of the study drug; The patients voluntarily participated in the study and signed the informed consent (or legal representative signed). It is expected that the patients have good compliance and can cooperate with the study according to the protocol requirements;

Exclusion Criteria:

1. Second-line or above chemotherapy or other anti-tumor drugs;
2. Cerebral edema requiring hormone dehydration treatment;
3. Major surgery performed within 4 weeks prior to the start of the study treatment or planned to be performed during the study program;
4. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as hepatitis B virus surface antigen [HBsAg] test positive, HBV-DNA ≥ 500 IU/ mL and abnormal liver function; Hepatitis C, defined as hepatitis C antibody [HCV-AB] positive, HCV-RNA higher than the lower limit of the assay and abnormal liver function) or co-infection with hepatitis B and hepatitis C;
5. The patient has an active bacterial or fungal infection (intravenous antibiotics are required at the beginning of the study);
6. Prior history of interstitial lung disease, drug-induced interstitial lung disease, radioactive pneumonia requiring steroid treatment, or any evidence of clinically active interstitial lung disease;
7. Arteriovenous thrombosis events, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, occurred within 6 months before enrollment;
8. A history of clinically significant cardiovascular disease, including but not limited to; (a) Congestive heart failure (NYHA grade > 2); (b) Unstable angina; (c) had a myocardial infarction within 3 months prior to signing the ICF; (d) Any supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
9. The average QTcF of three electrocardiograms was >470ms
10. Have had or had other systemic malignancies within the last 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ and ovarian cancer of the cervix);
11. a history of gastrointestinal diseases (such as Crohn's disease, ulcerative colitis, chronic diarrhea, and malabsorption) that affect the absorption of the test drug;
12. Use drugs or supplements known to be major contributors to CYP3A4.
13. known allergy to any test drug or its excipients;
14. Pregnancy, lactation patients, reproductive patients are unwilling to take effective contraceptive measures;
15. Prior use of CDK4/6 inhibitors;
16. Have a clear past history of neurological or psychiatric disorders, including epilepsy and dementia; Other conditions that the investigator deems inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer diagnosed by histopathology or cytology, TNM (8th) stage IV, accompanied by EGFR mutation, meningeal progression after previous platinum-containing two-drug chemotherapy and third-generation EGFR-TKI treatment, male and female, age ≥18 years, ECOG PS score 0-2
Sampling Method: Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
9 of participants | 1 year
  9 of participants

SECONDARY OUTCOMES:
ORR | 1 year
  Overall objective response rate
CNS PFS | 1 year
  CNS Progression-free survival
PFS | 1 year
  Progression-free survival
OS | through study completion, an average of 1 year
  Overall survival